CLINICAL TRIAL: NCT06946589
Title: Cardiac Changes After Effective Dose Carbetocin for Elective Caesarian Section
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jordan Leitch (Other)
Responsible Party: Sponsor-Investigator, Jordan Leitch, Dr. Jordan Leitch, Assistant Professor, Dept. of Anesthesiology/Critical Care, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69135
Record Dates: First submitted 2025-03-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Ischemia; Cesarian Section
Keywords: carbetocin; duratocin; cardiac symptoms
MeSH Terms: conditions — Coronary Artery Disease | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50mcg of Carbetocin (Experimental): Participants in this arm will receive 50mcg of carbetocin for post party hemorrhage prophylaxis at the the time of umbilical cord clamping during their cesarian section.
  Interventions: Drug: Carbetocin
- 100mcg of Carbetocin (Active Comparator): Participants in this arm will receive 100mcg of carbetocin for post party hemorrhage prophylaxis at the the time of umbilical cord clamping during their cesarian section.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — A uterotonic agent used for the prevention of postpartum hemorrhage in Cesarian section

SUMMARY:
The goal of this project is to examine the cardiac symptoms and physiologic changes after administration of a reduced dose of carbetocin in participants undergoing elective cesarian section.

* Does reduced dose carbetocin (50mcg) have fewer cardiac side effects than usual dose carbetocin (100mcg) when comparing patient reported symptoms, ECG changes and troponin increases?
* Is there a relationship between patient reported cardiac symptoms after carbetocin administration and subjective measures of cardiac ischemia (ECG changes and troponin increases? Researchers will compare 50mcg of carbetocin to the control group of 100mcg of carbetocin in patients undergoing elective cesarian section.

Participants will:

* Be given 50mcg or 100mcg of carbetocin during cesarian section
* Asked to report cardiac symptoms
* Be assessed for ECG changes and blood loss using standard of practice monitoring
* Have a troponin I blood test completed after delivery

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective cesarian section
* Primary and repeat cesarian section

Exclusion Criteria:

* Prior and current cardiovascular co-morbidities including pre-eclampsia
* BMI greater than 50
* Pre-existing bleeding disorders
* Allergy to carbetocin
* Age under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported symptoms | within 5 minutes of study drug administration
  Subjective patient reported symptoms of cardiac ischemia, reported with descriptive words

SECONDARY OUTCOMES:
Troponin I levels | One day after study drug administration
  Troponin I levels on blood work
ECG: ST segment | 5 minutes after study drug administration
  Changes to the ST segment on ECG

OTHER OUTCOMES:
Estimated blood loss during surgery | Within 1 hour of study drug administration
  Recorded from anesthesiologists assessment
Surgeons assessment of uterine tone | 3 minutes after study drug administration
  Assessed as a binary of adequate or not adequate
Hemoglobin change | Preoperatively and one day postoperatively
  Assessed as a difference between preoperative and postoperative hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Leitch, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No